CLINICAL TRIAL: NCT05289544
Title: Evaluating Alternative Delivery Models for Arthritis Self-management Interventions
Brief Title: Phone-Based Based Walk with Ease Program for Adults with Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00115106
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Arthritis; Gout; Fibromyalgia; Rheumatoid Arthritis; Osteoarthritis; Lupus Erythematosus, Systemic
Keywords: Arthritis; Physical activity; Intervention
MeSH Terms: conditions — Arthritis; Gout; Fibromyalgia; Arthritis, Rheumatoid; Osteoarthritis; Lupus Erythematosus, Systemic; Motor Activity | interventions — methyl hydroxyethyl cellulose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phone-Based Walk With Ease Program (Experimental): Telephone-based Walk With Ease Program adapted from the Arthritis Foundations program
  Interventions: Behavioral: Phone-Based Walk With Ease
- Delayed Phone-Based Walk With Ease Program (Other): Telephone-Based Walk With Ease Program starting after the 1 year assessment
  Interventions: Behavioral: Phone-Based Walk With Ease

INTERVENTIONS:
Behavioral: Phone-Based Walk With Ease — 6 week phone-delivered Walk With Ease Program

SUMMARY:
The objective of this study is to examine the short-term (6-weeks and 6 months) and long-term (1 year) effects of a phone-based version of Walk With Ease intervention.

DETAILED DESCRIPTION:
Participants will be randomized to either start the 6-week program immediately or after one year. Our Walk with Ease by Telephone (WWE-T) program is adapted from the original 6-week community-based group walking program developed by the Arthritis Foundation for adults with arthritis. The phone-based program will include 2 phone calls each week with a trained Walk With Ease Leader for 6 weeks. Assessments will be completed before at the start of the study, 6 weeks, 6 months and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* told by a doctor or other health professional that you have some form of arthritis, rheumatoid arthritis, gout, lupus, fibromyalgia
* able to read and write in English
* plan to live in the Columbia, SC region for next year
* willing to be randomized to either group
* complete all baseline measure

Exclusion Criteria:

* contraindications to exercise (besides arthritis)
* are pregnant, breastfeeding, or planning to become pregnant in the next year
* have a serious cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline to 6 weeks
  Visual analog scale (100 mm)
Change in pain | Baseline to 6 months
  Visual analog scale (100 mm)
Change in pain | Baseline to 12 months
  Visual analog scale (100 mm)
Change in physical function - chair stands | Baseline to 6 weeks
  repetitions completed during 30 second chair stand test
Change in physical function - chair stands | Baseline to 6 months
  repetitions completed during 30 second chair stand test
Change in physical function - chair stands | Baseline to 12 months
  repetitions completed during 30 second chair stand test
Change in physical function - 6 minute walk | Baseline to 6 weeks
  Distance walked (ft) during 6 minute walk test
Change in physical function - 6 minute walk | Baseline to 6 months
  Distance walked (ft) during 6 minute walk test
Change in physical function - 6 minute walk | Baseline to 12 months
  Distance walked (ft) during 6 minute walk test

SECONDARY OUTCOMES:
Change in Physical Limitations | Baseline to 6 weeks
  Health Assessment Questionnaire (HAQ) - Total score ranging from 0-3, with a higher score indicating more impairment or disability
Change in Physical Limitations | Baseline to 6 months
  Health Assessment Questionnaire (HAQ) - Total score ranging from 0-3, with a higher score indicating more impairment or disability
Change in Physical Limitations | Baseline to 12 months
  Health Assessment Questionnaire (HAQ) - Total score ranging from 0-3, with a higher score indicating more impairment or disability
Change in physical activity | Baseline to 6 weeks
  total moderate and vigorous intensity physical activity (>=2020 cpm) measured by Actigraph GT3x Link activity monitors
Change in physical activity | Baseline to 6 months
  total moderate and vigorous intensity physical activity (>=2020 cpm) measured by Actigraph GT3x Link activity monitors
Change in physical activity | Baseline to 12 months
  total moderate and vigorous intensity physical activity (>=2020 cpm) measured by Actigraph GT3x Link activity monitors
Change in arthritis management self-efficacy | Baseline to 6 weeks
  Confidence to manage symptoms of arthritis assessed by the Arthritis Self-Efficacy Scale. Total score 0-10 with higher scores indicating higher levels of self-efficacy for managing arthritis
Change in arthritis management self-efficacy | Baseline to 6 months
  Confidence to manage symptoms of arthritis assessed by the Arthritis Self-Efficacy Scale. Total score 0-10 with higher scores indicating higher levels of self-efficacy for managing arthritis
Change in arthritis management self-efficacy | Baseline to 12 months
  Confidence to manage symptoms of arthritis assessed by the Arthritis Self-Efficacy Scale. Total score 0-10 with higher scores indicating higher levels of self-efficacy for managing arthritis
Change in blood pressure | Baseline to 6 weeks
  Diastolic and systolic blood pressure measured in mmHg
Change in blood pressure | Baseline to 6 months
  Diastolic and systolic blood pressure measured in mmHg
Change in blood pressure | Baseline to 12 months
  Diastolic and systolic blood pressure measured in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available within 30 months of the completion of the project.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available within 30 months of the completion of the project.
Access Criteria: open access

REFERENCES:
- See also: Study Website — https://uofscwalkingstudy.com/